CLINICAL TRIAL: NCT01115933
Title: SPIRIT PRIME JAPAN (SV JAPAN)
Brief Title: A Clinical Evaluation of the XIENCE PRIME Small Vessel Everolimus Eluting Coronary Stent System in Japanese Population
Acronym: SV JAPAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-385
Record Dates: First submitted 2010-04-05; First posted 2010-05-04 (Estimated); Results first posted 2014-01-03 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-06

CONDITIONS: Vascular Disease; Myocardial Ischemia; Coronary Artery Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
Keywords: drug eluting stents; small vessel; Stents; Everolimus; Angioplasty
MeSH Terms: conditions — Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- XIENCE PRIME SV EECSS (Experimental): XIENCE PRIME SV EECSS: Small Vessel Everolimus Eluting Coronary Stent System
  Interventions: Device: XIENCE PRIME SV EECSS

INTERVENTIONS:
Device: XIENCE PRIME SV EECSS — Patients receiving XIENCE PRIME SV EECSS

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the AVJ-09-385 Small Vessel Everolimus Eluting Coronary Stent System (EECSS) (2.25 mm diameter stent) in treatment of subjects with ischemic heart disease caused by de novo lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 20 years of age.
2. Subject or a legally authorized representative must provide written informed consent prior to any study related procedure, per site requirements.
3. Subject must have evidence of myocardial ischemia (e.g., stable or unstable angina, silent ischemia, positive functional study or a reversible change in the electrocardiogram (ECG) consistent with ischemia).
4. Subject must be an acceptable candidate for coronary artery bypass graft (CABG) surgery.
5. Subject must agree to undergo all protocol-required follow-up procedures.
6. Subject must agree not to participate in any other clinical study for a period of one year following the index procedure.

Angiographic Inclusion Criteria

1. One (target) or two (one target and one non-target) de novo lesions each in a different epicardial vessel.
2. Lesion(s) must be located in a major artery or branch with a visually estimated diameter stenosis of ≥ 50% and < 100% with a TIMI flow of ≥ 1.
3. Lesion(s) must be located in a native coronary artery with reference vessel diameter (RVD) by visual estimation of ≥ 2.25 mm and < 2.5 mm.
4. Lesion(s) must be located in a native coronary artery with length by visual estimation of ≤ 22 mm.

Exclusion Criteria:

1. Subject has had a known diagnosis of acute myocardial infarction (AMI) preceding the index procedure (CK-MB ≥ 2 times upper limit of normal) and CK and CK-MB have not returned to within normal limits at the time of procedure.
2. The subject is currently experiencing clinical symptoms consistent with new onset AMI, such as nitrate-unresponsive prolonged chest pain with ischemic ECG changes.
3. Subject has current unstable cardiac arrhythmias associated with hemodynamic instability.
4. Subject has a known left ventricular ejection fraction (LVEF) < 40% (LVEF may be obtained at the time of the index procedure if the value is unknown and if necessary).
5. Subject has received coronary brachytherapy in any epicardial vessel.
6. Subject has received any organ transplant or is on a waiting list for any organ transplant.
7. Subject is receiving or scheduled to receive chemotherapy for malignancy within 30 days prior to or within one year after the index procedure.
8. Subject is receiving or scheduled to receive planned radiotherapy to the chest/mediastinum.
9. Subject is receiving immunosuppressant therapy or has known immunosuppressive or autoimmune disease (e.g. human immunodeficiency virus, systemic lupus erythematosus etc.).
10. Subject is receiving chronic anticoagulation therapy (e.g., heparin, warfarin).
11. Subject will require Low Molecular Weight Heparin (LMWH) post-procedure.
12. Subject has a known hypersensitivity or contraindication to aspirin, heparin, clopidogrel/ticlopidine, everolimus, cobalt, chromium, nickel, tungsten, acrylic and fluoro polymers or contrast sensitivity that cannot be adequately pre-medicated.
13. Elective surgery is planned within 6 months after the procedure that will require discontinuing either aspirin or clopidogrel.
14. Subject has a platelet count < 100,000 cells/mm3 or > 700,000 cells/mm3, a white blood cell (WBC) of < 3,000 cells/mm3, or documented or suspected liver disease (including laboratory evidence of hepatitis).
15. Subject has known renal insufficiency (examples being but not limited to serum creatinine level ≥ 2.0 mg/dL, or on dialysis).
16. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
17. Subject has had a cerebrovascular accident/stroke or transient ischemic neurological attack (TIA) within the past six months.
18. Subject has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has extensive peripheral vascular disease that precludes safe 5 French catheter insertion.
20. Subject has other medical illness (e.g., cancer) or known history of substance abuse (alcohol, cocaine, heroin etc.) that may cause non-compliance with the protocol, confound the data interpretation or is associated with a limited life expectancy (i.e., less than one year).
21. Subject is currently participating in another clinical study that has not yet completed its primary endpoint.
22. Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test*.

    * Whether a subject who met this criterion will be asked for pregnancy test will be decided per site standard. However, subject enrollment in the study is not allowed without pregnancy test result.

Angiographic Exclusion Criteria All angiographic exclusion criteria are based on visual estimation.

1. Target lesion located within an arterial or saphenous vein graft or distal to a diseased (vessel irregularity per angiogram and > 20% stenosed lesion) arterial or saphenous vein graft.
2. Target lesion involving a bifurcation with a side branch ≥ 2 mm in diameter and/or ostial lesion > 40% stenosed or side branch requiring protection guidewire, or side branch requiring dilatation.
3. Target lesion with total occlusion (TIMI flow 0), prior to crossing with the wire.
4. Another lesion requiring revascularization is located in the same epicardial vessel of the target lesion.
5. Restenotic lesion.
6. Aorto-ostial target lesion (within 3 mm of the aorta junction).
7. Lesion in the left main trunk (both target and non-target).
8. Lesion located within 2 mm of the origin of the LAD or LCX.
9. Extreme angulation (≥ 90 °) or excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion.
10. Heavy calcification proximal to or within the target lesion.
11. Target vessel contains thrombus as indicated in the angiographic images.
12. Target lesion has a high probability that a procedure other than pre-dilatation and stenting will be required at the time of index procedure for treatment of the target vessel (e.g. rotablator, DCA, cutting balloon).
13. Target vessel is previously treated* with any type of PCI (e.g. balloon angioplasty, stent, rotablator, DCA, cutting balloon) within 9 months of index procedure.
14. Non-target vessel was previously treated with any type of PCI within 90 days of index procedure.
15. Additional clinically significant lesion(s) in the target vessel or side branch for which PCI may be required within 90 days after the index procedure.

    * Target lesion must be separated ≥ 5 mm from a previously treated lesion (stenosis within 5 mm of previously treated lesion is regarded as "restenosis").

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takaaki Isshiki, MD, Principal Investigator — Teikyo University Hospital
Locations (14):
- Japan (14):
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Hokkaido Social Insurance Hospital Cardiovascular Center, Toyohira, Hokkaido
  - Teikyo University, Tokyo, Itabashi
  - Tokai University Hospital, Isehara, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Saiseikai Yokohama City Eastern Hospital, Yokohama, Kanagawa
  - Kumamoto Central Hospital, Kumamoto, Kumamoto
  - Kyoto University Hospital, Sakyo-ku, Kyoto
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nagoya Daini Red Cross Hospital, Shōwaku, Nagoya
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Sakurabashi Watanabe Hospital, Kita-ku, Osaka
  - Osaka University Hospital, Suita, Osaka
  - Tokushima Red Cross Hospital, Komatsushimachō, Tokushima

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 65 subjects at 15 Japanese sites were enrolled between April, 2010 and August, 2011.
Groups:
- XIENCE PRIME SV EECSS: XIENCE PRIME SV EECSS: XIENCE PRIME Small Vessel (2.25 mm) Everolimus Eluting Coronary Stent System
  XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
Period: Overall Study
Arm/Group | XIENCE PRIME SV EECSS
Started | 65
Completed | 64
Not Completed | 1
Not completed — Did not receive XIENCE PRIME SV | 1

BASELINE CHARACTERISTICS:
Population: Based on number of patients who received XIENCE PRIME SV EECSS
Groups:
- XIENCE PRIME SV EECSS: XIENCE PRIME SV Everolimus Eluting Coronary Stent System
  XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.63 (7.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 49
Region of Enrollment [Number; unit: participants]
  Japan | 64

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint of Cardiac Death/TV-MI/CI-TLR (TLF)
Description: Target lesion failure (TLF) is the composite of any of the following adverse events: Cardiac death, target vessel myocardial infarction (TV-MI) (per Protocol definition), Clinically indicated target lesion revascularization (CI-TLR)
Time Frame: 9 Months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

2. Secondary Outcome: Device Success (Lesion Based Analysis, Only for XIENCE PRIME SV)
Description: Device success is achievement final in-stent residual diameter stenosis of < 50% (by QCA). If adjunct treatment devices other than protocol defined device is used for target lesion treatment, malfunction of the investigational device occurring during the index procedure, are not regarded as device success. Use of a bail-out stent is still regarded as device success unless a device malfunction has occured. If QCA %DS is not available, the data is not included in analyses.
Time Frame: The period during an in-hospital stay of less than or equal to 7 days post index procedure.
Population: Intent to Treat Population (ITT)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 65
percentage of participants | 100.00 [94.48 to 100.00]

3. Secondary Outcome: Procedural Success(Subject Base Analysis)
Description: Procedure success is defined as achievement of a final in-stent diameter stenosis of < 50% (by QCA) using the investigational device (AVJ-09-385), without the occurrence MACE during the hospital stay (up to 7 days if a subject still in the hospital). If QCA %DS is not available, the data is not included in analyses.
Time Frame: The period during an in-hospital stay of less than or equal to 7 days post index procedure.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS: XIENCE PRIME SV EECSS EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 65
percentage of participants | 100.00 [94.48 to 100.00]

4. Secondary Outcome: Percent Diameter Stenosis (%DS), In-segment, In-stent, Proximal and Distal
Description: IN-STENT is defined as within the margins of the stent. IN-SEGMENT is defined as within the margins of the stent and 5 mm proximal and 5 mm distal to the stent.
  PROXIMAL is defined as within 5 mm of healthy tissue proximal to stent placement DISTAL is defined as within 5 mm of healthy tissue distal to stent placement
Time Frame: 8 months
Population: Full Analysis Set (FAS population)
Measure: Mean (Standard Deviation); unit: percentage of DS
Groups:
- XIENCE PRIME SV EECSS %DS In-segment; XIENCE PRIME SV EECSS %DS Distal: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS %DS In-stent; XIENCE PRIME SV EECSS %DS Proximal: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS %DS In-segment | XIENCE PRIME SV EECSS %DS In-stent | XIENCE PRIME SV EECSS %DS Proximal | XIENCE PRIME SV EECSS %DS Distal
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of DS | 19.80 (10.59) | 6.11 (11.65) | 12.32 (17.03) | 14.91 (8.12)

5. Secondary Outcome: Late Loss (LL), In-segment, In-stent, Proximal and Distal
Description: LATE LOSS (LL) calculated as MINIMUM LUMEN DIAMETER [MLD] post-procedure MINUS MLD at follow-up:
  In-segment Late Loss: in-segment MLD post-procedure - in segment MLD at follow-up In-stent Late Loss: in-stent MLD post-procedure - in-stent MLD at follow-up Proximal Late Loss: proximal MLD post-procedure - proximal MLD at follow-up (proximal defined as within 5 mm of healthy tissue proximal to stent placement) Distal Late Loss: distal MLD post-procedure - distal MLD at follow-up (distal defined as within 5 mm of healthy tissue distal to stent placement)
Time Frame: 8 months
Population: Full Analysis Set (FAS population)
Measure: Mean (Standard Deviation); unit: mm
Groups:
- XIENCE PRIME SV EECSS LL In-segment; XIENCE PRIME SV EECSS LL In-stent; XIENCE PRIME SV EECSS LL Distal: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS LL Proximal: XIENCE PRIME SV EECSS: Patients receivingXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS LL In-segment | XIENCE PRIME SV EECSS LL In-stent | XIENCE PRIME SV EECSS LL Proximal | XIENCE PRIME SV EECSS LL Distal
Number analyzed (Participants) | 64 | 64 | 64 | 64
mm | 0.12 (0.24) | 0.13 (0.25) | 0.08 (0.30) | 0.08 (0.25)

6. Secondary Outcome: Angiographic Binary Restenosis (ABR), In-segment, In-stent, Proximal and Distal
Description: as for outcome 4
Time Frame: 8 months
Population: Full Analysis Set (FAS population)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS ABR In-segment; XIENCE PRIME SV EECSS ABR In-stent; XIENCE PRIME SV EECSS ABR Proximal: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS ABR Distal: XIENCE PRIME SV EECSS : Patients receivingXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS ABR In-segment | XIENCE PRIME SV EECSS ABR In-stent | XIENCE PRIME SV EECSS ABR Proximal | XIENCE PRIME SV EECSS ABR Distal
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 4.8 [1.01 to 13.50] | 0 [0.00 to 5.78] | 3.7 [0.45 to 12.75] | 0 [0.00 to 6.38]

7. Secondary Outcome: Death (Cardiac, Vascular, Non-Cardiovascular, Per ARC Definition)
Description: DEATH (Per ARC Circulation 2007; 115: 2344-2351)
  All deaths are considered cardiac unless an unequivocal non-cardiac cause can be established. Specifically, any unexpected death even in patients with coexisting potentially fatal non-cardiac disease (e.g. cancer, infection) should be classified as cardiac.
Time Frame: 1 month
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - Cardiac: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - Vascular: XIENCE PRIME SV EECSS : Patients receiving AXIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - Non-Cardiovascular: XIENCE PRIME SV EECSS : Patients receivingXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - Cardiac | XIENCE PRIME SV EECSS - Vascular | XIENCE PRIME SV EECSS - Non-Cardiovascular
Number analyzed (Participants) | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00

8. Secondary Outcome: Death (Cardiac, Vascular, Non-Cardiovascular, Per ARC Definition)
Description: as for outcome 7
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - All Death Per ARC; XIENCE PRIME SV EECSS - Cardiac Death Per ARC; XIENCE PRIME SV EECSS - Vascular Death Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - Non-Cardiovascular Death Per ARC: XIENCE PRIME SV EECSS : Patients receiving AXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - All Death Per ARC | XIENCE PRIME SV EECSS - Cardiac Death Per ARC | XIENCE PRIME SV EECSS - Vascular Death Per ARC | XIENCE PRIME SV EECSS - Non-Cardiovascular Death Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 1.6 | 0.00 | 0.00 | 1.6

9. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions)
Description: Definitions in SPIRIT III Study:
  Q wave MI: Development of new, pathological Q wave on the ECG Non-Q wave MI: Elevation of CK levels to >=two times the upper limit of normal (ULN) with elevated CK-MB in the absence of new pathological Q waves Per ARC definition as published in 'Academic Research Consortium., Clinical end points in coronary stent trials: a case for standardized definitions.' Circulation 2007; 115: 2344-2351
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - QMI Per Protocol; XIENCE PRIME SV EECSS - NQMI Per Protocol; XIENCE PRIME SV EECSS - NQMI Per ARC Definitions: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - QMI Per ARC Definitions: XIENCE PRIME SV EECSS : Patients receivingXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - QMI Per Protocol | XIENCE PRIME SV EECSS - NQMI Per Protocol | XIENCE PRIME SV EECSS - QMI Per ARC Definitions | XIENCE PRIME SV EECSS - NQMI Per ARC Definitions
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00 | 0.00

10. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions)
Description: as for outcome 9
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - NQMI Per Protocol: XIENCE PRIME SV EECSS : Patients receivingXIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - QMI Per ARC: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - NQMI Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - QMI Per Protocol | XIENCE PRIME SV EECSS - NQMI Per Protocol | XIENCE PRIME SV EECSS - QMI Per ARC | XIENCE PRIME SV EECSS - NQMI Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00 | 0.00

11. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions) Attributable to Target Vessel (TV-MI)
Description: as for outcome 9
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS- TV-QMI Per Protocol; XIENCE PRIME SV EECSS - TV-NQMI Per Protocol; XIENCE PRIME SV EECSS - TV-QMI Per ARC; XIENCE PRIME SV EECSS - TV-NQMI Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS- TV-QMI Per Protocol | XIENCE PRIME SV EECSS - TV-NQMI Per Protocol | XIENCE PRIME SV EECSS - TV-QMI Per ARC | XIENCE PRIME SV EECSS - TV-NQMI Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00 | 0.00

12. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions) Attributable to Target Vessel (TV-MI)
Description: as for outcome 9
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - TV-QMI Per Protocol; XIENCE PRIME SV EECSS - TV-NQMI Per Protocol; XIENCE PRIME SV EECSS - TV-QMI Per ARC; XIENCE PRIME SV EECSS - TV-NQMI Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - TV-QMI Per Protocol | XIENCE PRIME SV EECSS - TV-NQMI Per Protocol | XIENCE PRIME SV EECSS - TV-QMI Per ARC | XIENCE PRIME SV EECSS - TV-NQMI Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00 | 0.00

13. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions) Not Attributable to Target Vessel (NTV-MI)
Description: as for outcome 9
Time Frame: 1 month
Population: FAS Population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS Non-Target Vessel QMI Per Protocol; XIENCE PRIME SV EECSS Non-Target Vessel NQMI Per Protocol; XIENCE PRIME SV EECSS Non-Target Vessel QMI Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS Non-Target Vessel NQMI Per ARC: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS Non-Target Vessel QMI Per Protocol | XIENCE PRIME SV EECSS Non-Target Vessel NQMI Per Protocol | XIENCE PRIME SV EECSS Non-Target Vessel QMI Per ARC | XIENCE PRIME SV EECSS Non-Target Vessel NQMI Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0 | 0 | 0 | 0

14. Secondary Outcome: Myocardial Infarction (MI: QMI and NQMI, Both Per SPIRIT III Protocol and Per ARC Definitions) Not Attributable to Target Vessel (NTV-MI)
Description: as for outcome 9
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - NTV-QMI Per Protocol; XIENCE PRIME SV EECSS - NTV-QMI Per ARC; XIENCE PRIME SV EECSS - NTV-NQMI Per ARC: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - NTV-NQMI Per Protocol: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - NTV-QMI Per Protocol | XIENCE PRIME SV EECSS - NTV-NQMI Per Protocol | XIENCE PRIME SV EECSS - NTV-QMI Per ARC | XIENCE PRIME SV EECSS - NTV-NQMI Per ARC
Number analyzed (Participants) | 64 | 64 | 64 | 64
percentage of participants | 0.00 | 0.00 | 0.00 | 0.00

15. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition)
Description: Any revascularization for in-segment restenosis will be considered TLR."Segment" is defined as the area within the margins of the stent and 5 mm proximal and 5 mm distal to the stent. Revascularization was considered clinically indicated if there was >70% diameter stenosis on angiography or >50% stenosis together with a positive stress test or ischaemic symptoms.
Time Frame: 1 month
Population: Full analysis set (FAS) population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

16. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition)
Description: Any revascularization for in-segment restenosis will be considered TLR. "Segment" is defined as the area within the margins of the stent and 5 mm proximal and 5 mm distal to the stent. Revascularization was considered clinically indicated if there was >70% diameter stenosis on angiography or >50% stenosis together with a positive stress test or ischaemic symptoms.
Time Frame: 9 months
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 3.1

17. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition) Clinically-indicated TLR (CI-TLR)
Description: as for outcome 16
Time Frame: 1 month
Population: Full analysis set (FAS) population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

18. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition) Clinically-indicated TLR (CI-TLR)
Description: as for outcome 16
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

19. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition) Not Clinically-indicated TLR (NCI-TLR)
Description: as for outcome 16
Time Frame: 1 month
Population: Full analysis set (FAS) population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

20. Secondary Outcome: Target Lesion Revascularization (TLR, Per ARC Definition) Not Clinically-indicated TLR (NCI-TLR)
Description: as for outcome 16
Time Frame: 9 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 3.1

21. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself. Revascularization was considered clinically indicated if there was >70% diameter stenosis on angiography or >50% stenosis together with a positive stress test or ischaemic symptoms.
Time Frame: 1 month
Population: FAS Population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0

22. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition)
Description: as for outcome 21
Time Frame: 9 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 3.1

23. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition) Clinically-indicated TVR (CI-TVR)
Description: as for outcome 21
Time Frame: 1 month
Population: Full analysis set (FAS) population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

24. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition) Clinically-indicated TVR (CI-TVR)
Description: as for outcome 21
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 1.6

25. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition) Not Clinically-indicated TVR (NCI-TVR)
Description: as for outcome 21
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

26. Secondary Outcome: Target Vessel Revascularization (TVR, Per ARC Definition) Not Clinically-indicated TVR (NCI-TVR)
Description: as for outcome 21
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 3.1

27. Secondary Outcome: Composite Endpoint of Cardiac Death/All MI
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

28. Secondary Outcome: Composite Endpoint of Cardiac Death/All MI
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.0

29. Secondary Outcome: Composite Endpoint of All Death/All MI/All Revascularization (DMR)
Description: DMR event (all death, all MI (per protocol or per ARC), all revascularization, respectively).
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

30. Secondary Outcome: Composite Endpoint of All Death/All MI/All Revascularization (DMR)
Description: DMR event (all death, all MI (per protocol or per ARC), all revascularization, respectively).
Time Frame: 9 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 10.9

31. Secondary Outcome: Composite Endpoint of Cardiac Death/TV-MI/CI-TLR (TLF)
Description: Target lesion failure (TLF) is defined as a composite of cardiac death, target-vessel related myocardial infarction (TV-MI) and clinically-indicated target lesion revascularization (CI-TLR).
Time Frame: 1 month
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

32. Secondary Outcome: Composite Endpoint of Cardiac Death/All MI/CI-TLR (MACE)
Description: Major adverse cardiac events (MACE) is defined as the composite of cardiac death, all myocardial-infarction, and clinically-indicated target lesion revascularization (CI-TLR).
Time Frame: 1 month
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

33. Secondary Outcome: Composite Endpoint of Cardiac Death, All MI and CI-TLR (MACE)
Description: as for outcome 32
Time Frame: 9 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.0

34. Secondary Outcome: All Coronary Revascularization
Time Frame: 1 months
Population: Full Analysis Set (FAS population)
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.00

35. Secondary Outcome: All Coronary Revascularization
Time Frame: 9 months
Population: FAS population
Measure: Number; unit: percentage of participants
Arm/Group | XIENCE PRIME SV EECSS
Number analyzed (Participants) | 64
percentage of participants | 0.0

36. Secondary Outcome: Acute Stent Thrombosis
Description: Stent thrombosis (ST) was defined according to the ARC guidelines as follows: definite: acute coronary syndrome and angiographic or pathological confirmation of ST; probable: unexplained death ≤30 days or target vessel MI without angiographic information; and possible: unexplained death >30 days after stent placement."
Time Frame: <24 hours
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - ST Definite; XIENCE PRIME SV EECSS - ST Possible; XIENCE PRIME SV EECSS - ST Definite/Probable: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - ST Probable: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - ST Definite/Probable/Possible: XIENCE PRIME SV EECSS : Patients receivingXIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - ST Definite | XIENCE PRIME SV EECSS - ST Probable | XIENCE PRIME SV EECSS - ST Possible | XIENCE PRIME SV EECSS - ST Definite/Probable | XIENCE PRIME SV EECSS - ST Definite/Probable/Possible
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

37. Secondary Outcome: Subacute Stent Thrombosis
Description: Stent thrombosis was defined according to the ARC guidelines as follows: definite: acute coronary syndrome and angiographic or pathological confirmation of ST; probable: unexplained death ≤30 days or target vessel MI without angiographic information; and possible: unexplained death >30 days after stent placement."
Time Frame: 1-30 days
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - ST Possible: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - ST Definite/Probable/Possible: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - ST Definite | XIENCE PRIME SV EECSS - ST Probable | XIENCE PRIME SV EECSS - ST Possible | XIENCE PRIME SV EECSS - ST Definite/Probable | XIENCE PRIME SV EECSS - ST Definite/Probable/Possible
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

38. Secondary Outcome: Acute/Subacute Stent Thrombosis
Description: as for outcome 37
Time Frame: 0-30 days
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - ST Definite; XIENCE PRIME SV EECSS - ST Possible; XIENCE PRIME SV EECSS - ST Definite/Probable/Possible: XIENCE PRIME SV EECSS: Patients receiving XIENCE PRIME SV EECSS
- XIENCE PRIME SV EECSS - ST Probable; XIENCE PRIME SV EECSS - ST Definite/Probable: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - ST Definite | XIENCE PRIME SV EECSS - ST Probable | XIENCE PRIME SV EECSS - ST Possible | XIENCE PRIME SV EECSS - ST Definite/Probable | XIENCE PRIME SV EECSS - ST Definite/Probable/Possible
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
percentage of participants | 0.0 | 0.0 | 0.00 | 0.00 | 0.0

39. Secondary Outcome: Late Stent Thrombosis
Description: as for outcome 37
Time Frame: 31 - 298 days
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS- ST Probable; XIENCE PRIME SV EECSS - ST Possible; XIENCE PRIME SV EECSS - ST Definite/Probable; XIENCE PRIME SV EECSS - ST Definite/Probable/Possible: XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - ST Definite | XIENCE PRIME SV EECSS- ST Probable | XIENCE PRIME SV EECSS - ST Possible | XIENCE PRIME SV EECSS - ST Definite/Probable | XIENCE PRIME SV EECSS - ST Definite/Probable/Possible
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

40. Secondary Outcome: Overall Stent Thrombosis
Description: as for outcome 37
Time Frame: 0 - 298 days
Population: FAS population
Measure: Number; unit: percentage of participants
Groups:
- XIENCE PRIME SV EECSS - ST Possible: XIENCE PRIME SV EECSS: Small Vessel Everolimus Eluting Coronary Stent System
  XIENCE PRIME SV EECSS : Patients receiving XIENCE PRIME SV EECSS
Arm/Group | XIENCE PRIME SV EECSS - ST Definite | XIENCE PRIME SV EECSS - ST Probable | XIENCE PRIME SV EECSS - ST Possible | XIENCE PRIME SV EECSS - ST Definite/Probable | XIENCE PRIME SV EECSS - ST Definite/Probable/Possible
Number analyzed (Participants) | 64 | 64 | 64 | 64 | 64
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Nine (9) month post procedure data which includes events which occurred up to 298 days.
Groups:
- AVJ-09-385 SV EECSS: SV EECSS: Small Vessel Everolimus Eluting Coronary Stent System
  AVJ-09-385 EECSS : Patients receiving AVJ-09-385 EECSS
Arm/Group | AVJ-09-385 SV EECSS
Serious Adverse Events (participants affected / at risk) | 10/64
Other Adverse Events (participants affected / at risk) | 4/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVJ-09-385 SV EECSS (N=64)
Angina unstable (Cardiac disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2)
(Eye disorders) | 1 (1)
(Infections and infestations) | 1 (1)
(Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVJ-09-385 SV EECSS (N=64)
hordeolum, influenza, nasopharyngitis (Infections and infestations) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days